CLINICAL TRIAL: NCT02227992
Title: A Prospective, Randomized, Controlled, Study Evaluating the Safety and Effectiveness of EVARREST® Sealant Matrix in Controlling Mild or Moderate Hepatic Parenchyma or Soft Tissue Bleeding During Open Abdominal, Retroperitoneal, Pelvic and Thoracic (Non-cardiac) Surgery in Paediatric Patients
Brief Title: The EVARREST® Paediatric Mild/Moderate Liver and Soft Tissue Bleeding Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 400-12-004; 2013-003557-24 (EudraCT Number)
Record Dates: First submitted 2014-07-28; First posted 2014-08-28 (Estimated); Results first posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2022-10

CONDITIONS: Hemorrhage; Soft Tissue Bleeding; Hepatic Parenchyma Bleeding
Keywords: Fibrin Sealant; Hemostatics; Coagulants
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EVARREST™ Sealant Matrix (Experimental): EVARREST™ Sealant Matrix/Fibrin Sealant Patch is a sterile bio-absorbable combination product consisting of two constituent parts- a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin).
  Interventions: Biological: EVARREST™ Sealant Matrix
- SURGICEL® Absorbable Hemostat (Active Comparator): SURGICEL® Absorbable Hemostat (oxidized regenerated cellulose) is a sterile absorbable knitted fabric prepared by the controlled oxidation of regenerated cellulose.
  Interventions: Device: SURGICEL®

INTERVENTIONS:
Biological: EVARREST™ Sealant Matrix — EVARREST® Fibrin Sealant Patch is a sterile, bio-absorbable combination product, comprised of two biological components (human plasma-derived fibrinogen and thrombin) embedded in a flexible composite patch component.
  Other Names: EVARREST™ Fibrin Sealant Patch
  Arms: EVARREST™ Sealant Matrix
Device: SURGICEL® — SURGICEL® Absorbable Hemostat is a sterile absorbable knitted fabric prepared by the controlled oxidation of regenerated cellulose.
  Other Names: oxidized regenerated cellulose
  Arms: SURGICEL® Absorbable Hemostat

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of EVARREST™ Sealant Matrix (EVARREST™ Fibrin Sealant Patch) (EVARREST™) in controlling mild or moderate soft tissue & parenchymal bleeding during open hepatic, abdominal, pelvic, retroperitoneal, and thoracic (non-cardiac) surgery in paediatric patients.

DETAILED DESCRIPTION:
This is an open label, prospective, randomised, multicentre, controlled, clinical study comparing EVARREST to SURGICEL (oxidized regenerated cellulose (ORC)) (Control) as an adjunct to haemostasis when conventional methods of controlling mild or moderate bleeding are ineffective or impractical during surgery in paediatric patients.

At least 40 qualified paediatric subjects with an appropriate mild or moderate bleeding Target Bleeding Site (TBS) will be randomised in a 1:1 allocation ratio to either EVARREST or SURGICEL (control). Absolute time to haemostasis will be assessed as well as haemostasis at 4 and 10 minutes from randomisation.

Enrolment will be staggered by age (as required by the European Medicines Agency (EMA) Paediatric Committee). The first 36 subjects enrolled will be aged ≥1 years to <18 years of age. Enrolment of a subsequent group will include 4 subjects from 1 month (≥ 28 days from birth) to <1 year of age will follow. Ongoing safety assessment will ensure adequate safety monitoring occur during the staged enrolment.

Subjects will be followed post-operatively through hospital discharge and at 30 days (+/-14 days) post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric subjects aged ≥28 days (≥ 1 month) to <18 years, requiring non-emergent open hepatic, abdominal, retroperitoneal, pelvic or thoracic (non-cardiac) surgical procedures. i) The first 36 subjects to be enrolled will be subjects aged ≥1 years to <18 years. ii) The next 4 subjects to be enrolled will be subjects aged ≥28 days to <1 year.
* The subject's parent/legal guardian must be willing to give permission for the subject to participate in the trial, and provide written informed consent for the subject. In addition, assent must be obtained from paediatric subjects who possess the intellectual and emotional ability to comprehend the concepts involved in the trial. If the paediatric subject is not able to provide assent (due to age, maturity and/or inability to intellectually and/or emotionally comprehend the trial), the parent/legal guardian's written Informed Consent for the subject will be acceptable for the subject to be included in the study.
* Presence of an appropriate mild or moderate bleeding soft tissue or hepatic parenchyma Target Bleeding Site (TBS) identified intra-operatively by the surgeon;
* Ability to firmly press trial treatment at TBS until 4 minutes after randomisation

Exclusion Criteria:

* Subjects with known intolerance to blood products or to one of the components of the study product or is unwilling to receive blood products;
* Female subjects, who are of childbearing age (i.e. adolescent), who are pregnant or nursing;
* Subject is currently participating or plans to participate in any other investigational device or drug without prior approval from the Sponsor;
* Subjects who are known, current alcohol and/or drug abusers
* Subjects admitted for trauma surgery
* Subjects with any pre or intra-operative findings identified by the surgeon that may preclude conduct of the study procedure.
* Subject with TBS in an actively infected field (Class III Contaminated or Class IV Dirty or Infected)
* TBS is from large defects in arteries or veins where the injured vascular wall requires repair with maintenance of vessel patency and which would result in persistent exposure of the EVARREST™ or SURGICEL® to blood flow and pressure during healing and absorption of the product;
* TBS with major arterial bleeding requiring suture or mechanical ligation;
* Bleeding site is in, around, or in proximity to foramina in bone, or areas of bony confine.

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kocharian, MD, PhD, Study Director — Ethicon, Inc.
Locations (10):
- Belgium (3):
  - Clinical Investigation Site #32, Brussels
  - Investigative Site #30, Genk
  - Clinical Investigation Site #31, Ghent
- United Kingdom (7):
  - Clinical Investigation Site #21, Birmingham
  - Clinical Investigation Site #22, Leeds
  - Clinical Investigation Site #20, Liverpool
  - Clinical Investigation Site #26, London
  - Clinical Investigation Site #23, London
  - Clinical Investigation Site #25, Nottingham
  - Clinical Investigation Site #24, Southampton

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- EVARREST Sealant Matrix: Participants with mild or moderate target bleeding site (TBS) were treated with EVARREST which was applied immediately to the actively bleeding TBS. EVARREST Sealant Matrix/Fibrin Sealant Patch was a sterile bio-absorbable combination product consisting of two constituent parts a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin).
- SURGICEL Absorbable Hemostat (Control): Participants with mild or moderate TBS were treated with SURGICEL which was applied immediately to the actively bleeding TBS. SURGICEL Absorbable Hemostat (oxidized regenerated cellulose) was a sterile absorbable knitted fabric prepared by the controlled oxidation of regenerated cellulose.
Period: Overall Study
Arm/Group | EVARREST Sealant Matrix | SURGICEL Absorbable Hemostat (Control)
Started | 20 | 20
Completed | 19 | 19
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EVARREST Sealant Matrix | SURGICEL Absorbable Hemostat (Control) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Full Range); unit: years] | 3.0 [0.8 to 13.0] | 4.0 [0.3 to 14.0] | 3.0 [0.3 to 14.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 19 | 18 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 18 | 17 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Absolute Time to Haemostasis (TTH)
Description: Absolute TTH, defined as the absolute time elapsed from randomization to the last moment in time at which detectable bleeding at the target bleeding site (TBS) was observed.
Time Frame: Up to 1 day (Intraoperative)
Population: The Full Analysis Set (FAS; equivalent to the Intent-to-Treat [ITT] set) consisted of all randomized participants. Participants who did not complete the procedure with the use of EVARREST or SURGICEL after randomization were included in the FAS analysis.
Measure: Median (Full Range); unit: Minutes
Arm/Group | EVARREST Sealant Matrix | SURGICEL Absorbable Hemostat (Control)
Number analyzed (Participants) | 20 | 20
Minutes | 4.0 [4.0 to 117.0] | 4.0 [4.0 to 39.0]

2. Secondary Outcome: Percentage of Participants Achieving Haemostatic Success at 4 Minutes Following Randomization With No Bleeding Requiring Treatment at the Target Bleeding Site Occurring Any Time Prior to Final Fascial Closure
Description: Percentage of participants achieving haemostatic success at 4 minutes following randomization with no bleeding requiring treatment at the TBS occurring any time prior to final fascial closure were reported.
Time Frame: 4 minutes post randomization (up to 1 day; intraoperative)
Population: The FAS (equivalent to the ITT set) consisted of all randomized participants. Participants who did not complete the procedure with the use of EVARREST or SURGICEL after randomization were included in the FAS analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | EVARREST Sealant Matrix | SURGICEL Absorbable Hemostat (Control)
Number analyzed (Participants) | 20 | 20
Percentage of Participants | 80.0 [56.3 to 94.3] | 60.0 [36.1 to 80.9]

3. Secondary Outcome: Percentage of Participants Achieving Haemostatic Success at 10 Minutes Following Randomization With No Bleeding Requiring Treatment at the Target Bleeding Site Occurring Any Time Prior to Final Fascial Closure
Description: Percentage of participants achieving haemostatic success at 10 minutes following randomization with no bleeding requiring treatment at the TBS occurring any time prior to final fascial closure were reported.
Time Frame: 10 minutes post randomization (up to 1 day; intraoperative)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | EVARREST Sealant Matrix | SURGICEL Absorbable Hemostat (Control)
Number analyzed (Participants) | 20 | 20
Percentage of Participants | 95.0 [75.1 to 99.9] | 90.0 [68.3 to 98.8]

4. Secondary Outcome: Percentage of Participants With No Re-bleeding at the Target Bleeding Site
Description: Percentage of participants with no re-bleeding at the TBS were reported.
Time Frame: Up to 44 days post-surgery on Day 0
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | EVARREST Sealant Matrix | SURGICEL Absorbable Hemostat (Control)
Number analyzed (Participants) | 20 | 20
Percentage of Participants | 95.0 | 85.0

5. Secondary Outcome: Number of Participants With Adverse Events (AEs) That Were Potentially Related To Bleeding at the TBS
Description: Number of participants With AEs that were potentially related to bleeding at the TBS were reported. An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time Frame: Up to 44 days post-surgery on Day 0
Population: The safety analysis set consists of all participants who received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | EVARREST Sealant Matrix | SURGICEL Absorbable Hemostat (Control)
Number analyzed (Participants) | 20 | 20
Participants | 1 | 3

6. Secondary Outcome: Number of Participants With AEs That Were Potentially Related To Thrombotic Events
Description: Number of participants with AEs that were potentially related to thrombotic events (sponsor assessment) were reported. An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time Frame: Up to 44 days post-surgery on Day 0
Population: The safety analysis set consists of all participants who received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | EVARREST Sealant Matrix | SURGICEL Absorbable Hemostat (Control)
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

7. Secondary Outcome: Number of Participants Who Required Re-treatment At The Target Bleeding Site
Description: Number of participants who required re-treatment at the TBS were reported.
Time Frame: Up to 44 days post-surgery on Day 0
Population: The safety analysis set consists of all participants who received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | EVARREST Sealant Matrix | SURGICEL Absorbable Hemostat (Control)
Number analyzed (Participants) | 20 | 20
Participants | 1 | 5

8. Secondary Outcome: Number of Participants With Adverse Events
Description: An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time Frame: Up to 44 days post-surgery on Day 0
Population: The safety analysis set consists of all participants who received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | EVARREST Sealant Matrix | SURGICEL Absorbable Hemostat (Control)
Number analyzed (Participants) | 20 | 20
Participants | 18 | 18

9. Secondary Outcome: Change From Baseline to Post-surgery in Haemoglobin
Description: Change from baseline to post-surgery in haemoglobin were reported.
Time Frame: From baseline up to hospital discharge (up to Day 44 post-surgery on Day 0)
Population: The safety analysis set consists of all participants who received treatment. Here, 'N' (number of participants analyzed) signifies number of participants who were analyzed for this outcome measure.
Measure: Median (Full Range); unit: grams/liter (g/L)
Arm/Group | EVARREST Sealant Matrix | SURGICEL Absorbable Hemostat (Control)
Number analyzed (Participants) | 19 | 20
grams/liter (g/L) | 0.0 [-56.0 to 43.0] | -10.0 [-150.0 to 44.0]

10. Secondary Outcome: Change From Baseline to Post-surgery in Haematocrit
Description: Change from baseline to post-surgery in Haematocrit was reported.
Time Frame: From baseline up to hospital discharge (up to Day 44 post-surgery on Day 0)
Population: as for outcome 9
Measure: Median (Full Range); unit: Liter of cells per liter of blood (L/L)
Arm/Group | EVARREST Sealant Matrix | SURGICEL Absorbable Hemostat (Control)
Number analyzed (Participants) | 19 | 20
Liter of cells per liter of blood (L/L) | 0.0 [-0.2 to 0.1] | -0.0 [-0.1 to 0.1]

11. Secondary Outcome: Change From Baseline to Post-surgery in Platelet Count
Description: Change from baseline to post-surgery in platelet count was reported.
Time Frame: From baseline up to hospital discharge (up to Day 44 post-surgery on Day 0)
Population: as for outcome 9
Measure: Median (Full Range); unit: 10^9 cells per liter
Arm/Group | EVARREST Sealant Matrix | SURGICEL Absorbable Hemostat (Control)
Number analyzed (Participants) | 19 | 20
10^9 cells per liter | -89.0 [-531.0 to 112.0] | -71.5 [-259.0 to 386.0]

12. Secondary Outcome: Estimated Volume of Blood Loss
Description: Estimated volume of intra-operative blood loss (including but not limited to the TBS) was reported.
Time Frame: Up to 1 day (intraoperative)
Population: The FAS consisted of all randomized participants. Participants who did not completed the procedure with the use of EVARREST or SURGICEL after randomization were included in the FAS analysis.
Measure: Median (Full Range); unit: Milliliter (mL)
Arm/Group | EVARREST Sealant Matrix | SURGICEL Absorbable Hemostat (Control)
Number analyzed (Participants) | 20 | 20
Milliliter (mL) | 100.0 (0.0) [0.0 to 800.0] | 200.0 (15.0) [15.0 to 2000.0]

13. Secondary Outcome: Number of Participants Who Received Blood Transfusions
Description: Number of participants who received blood transfusions (red blood cells [RBCs], whole blood, fresh frozen plasma, platelets, and cryoprecipitates) were reported.
Time Frame: Up to 44 days post-surgery on Day 0
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | EVARREST Sealant Matrix | SURGICEL Absorbable Hemostat (Control)
Number analyzed (Participants) | 12 | 11
Participants
  Packed RBCs (0 Unit) | 3 | 2
  Packed RBCs (1 Unit) | 4 | 4
  Packed RBCs (2 Units) | 4 | 3
  Packed RBCs (3 Units) | 1 | 1
  Packed RBCs (6 Units) | 0 | 1
  Whole Blood (0 Unit) | 9 | 9
  Whole Blood (1 Unit) | 2 | 1
  Whole Blood (2 Units) | 1 | 1
  Fresh Frozen Plasma (0 Unit) | 10 | 11
  Fresh Frozen Plasma (2 Units) | 1 | 0
  Fresh Frozen Plasma (5 Units) | 1 | 0
  Platelets (0 Units) | 8 | 9
  Platelets (1 Unit) | 3 | 1
  Platelets (2 Units) | 1 | 0
  Platelets (3 Units) | 0 | 1
  Cryoprecipitates (0 Units) | 12 | 11

14. Primary Outcome: Absolute Time to Haemostasis (TTH) by Age Group
Description: Absolute TTH, defined as the absolute time elapsed from randomization to the last moment in time at which detectable bleeding at the TBS was observed.
Time Frame: Up to 1 day (Intraoperative)
Population: The Full Analysis Set (FAS; equivalent to the ITT set) consisted of all randomized participants. Participants who did not complete the procedure with the use of EVARREST or SURGICEL after randomization were included in the FAS analysis. Here 'n' (number analyzed) signifies number of participants analyzed for specified categories.
Measure: Median (Full Range); unit: Minutes
Arm/Group | EVARREST Sealant Matrix | SURGICEL Absorbable Hemostat (Control)
Number analyzed (Participants) | 20 | 20
Minutes
  Infants and toddlers (28 days to less than 24 months): number analyzed (Participants) | 6 | 5
  Infants and toddlers (28 days to less than 24 months) | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 6.9]
  Children (2 to 11 years): number analyzed (Participants) | 11 | 11
  Children (2 to 11 years) | 4.0 [4.0 to 117.0] | 4.0 [4.0 to 39.0]
  Adolescent (12 to less than 18 years): number analyzed (Participants) | 3 | 4
  Adolescent (12 to less than 18 years) | 4.0 [4.0 to 7.5] | 4.0 [4.0 to 10.0]

ADVERSE EVENTS:
Time Frame: Up to 44 days post-surgery on Day 0
Description: The safety analysis set consists of all participants who received treatment.
Arm/Group | EVARREST Sealant Matrix | SURGICEL Absorbable Hemostat (Control)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 4/20 | 5/20
Other Adverse Events (participants affected / at risk) | 18/20 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVARREST Sealant Matrix (N=20) | SURGICEL Absorbable Hemostat (Control) (N=20)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Bloody Discharge (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVARREST Sealant Matrix (N=20) | SURGICEL Absorbable Hemostat (Control) (N=20)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 3 (3)
Tachycardia (Cardiac disorders) | 10 (10) | 7 (9)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (7) | 6 (7)
Haemorrhage (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0)
Puncture site discharge (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 9 (10)
Procedural hypotention (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 7 (7)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood alkaline phosphate decreased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2) | 2 (2)
International normalized ratio increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 2 (2)
Urine output decreased (Investigations) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Horner's syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Vulval oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Device occlusion (General disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 2 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Joint instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Anal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication or other public presentation of results from this study requires prior review by ETHICON. Draft abstracts, manuscripts, and materials for presentation at scientific meetings must be sent to the sponsor at least 60 days prior to submission for publication, public dissemination, or review by a publication committee.

DOCUMENTS (2):
  • Study Protocol (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT02227992/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT02227992/SAP_001.pdf